CLINICAL TRIAL: NCT01217541
Title: Collaboration Between Department of Old Age Psychiatry and Nursing Homes
Acronym: SAM-AKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Helse Sor-Ost (Other Government); Norwegian Department of Health and Social Affairs (Other Government)
Responsible Party: Principal Investigator, Sverre Bergh, Research Director Centre for Old Age Psychiatric Research, Sykehuset Innlandet HF
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 50022
Record Dates: First submitted 2010-09-22; First posted 2010-10-08 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Dementia; Alzheimer's Disease; Behavioral Symptoms; Agitation
Keywords: Dementia; BPSD; Quality of Life; Person-centred care; Job satisfaction; Nursing home; Primary care
MeSH Terms: conditions — Dementia; Alzheimer Disease; Behavioral Symptoms; Psychomotor Agitation | interventions — Educational Status; Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education and supervision (Other): Personnel in nursing home units get intervention in form of education and supervision
  Interventions: Other: Education and Supervision; Other: Control
- Control (No Intervention): Only registering of patient and personnel data in the beginning and the end of the study without any form of intervention.

INTERVENTIONS:
Other: Education and Supervision — Implementation of Scales in the care of patients with dementia in nursing home units with focus on person-centred care. Supervision of caregivers on a regular basis.
  Other Names: Departments in NHs that do not get any intervention.
  Arms: Education and supervision
Other: Control — A control group of nursing home units that do not get any form of active intervention
  Other Names: Education; Supervision
  Arms: Education and supervision

SUMMARY:
Dementia is a serious health problem showing an increasing prevalence rate with increasing age. In Norway, about 80% of nursing home patients have dementia. The mean age of nursing home residents in Norway is around 84 years. Disruptive and agitated behaviour affect 30-50% of all individuals with dementia at some point in the course of the illness. In addition, they have a combination of physical and psychological diseases which necessitates a close collaboration between different specialities in medicine and Old Age psychiatry. In collaboration with the communalities, our Old Age psychiatry services want to provide a new approach to this challenge and validate it on patient and personnel level.

ELIGIBILITY:
Inclusion Criteria:

* All patients at nursing home units

Exclusion Criteria:

* Patients that are in a final state and patients that have not been at the nursing home unit more than two weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Quality of Life in Severe Dementia (QUALID), Person-Centred Care Assessment Tool (P-CAT, 2010) | 12 months after baseline assessment
  Evaluate a new model of collaboration between a specialized department of Old Age Psychiatry and nursing home units to optimize patient care and job satisfaction of the caregivers.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory - Nursing Home version, Cornell Scale of Depression in Dementia, Registration of Constraints (Kirkevold, 2004) | 12 months after baseline assessment
  In addition, we want to carry out a qualitative evaluation of the process of implementation of new scales and the effect of supervision on personnel and patients

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbæk, PhD, Principal Investigator — Sykehuset Innlandet HF
Locations (1):
- Lillehammer sykehjem, Lillehammer, Oppland, Norway

REFERENCES:
- [Background] Selbaek G, Kirkevold O, Engedal K. Psychiatric and behavioural symptoms and the use of psychotropic medication in Special Care Units and Regular Units in Norwegian nursing homes. Scand J Caring Sci. 2008 Dec;22(4):568-73. doi: 10.1111/j.1471-6712.2007.00576.x. Epub 2008 Sep 16. PMID 18801019
- [Background] Kirkevold O, Laake K, Engedal K. Use of constraints and surveillance in Norwegian wards for the elderly. Int J Geriatr Psychiatry. 2003 Jun;18(6):491-7. doi: 10.1002/gps.883. PMID 12789669